CLINICAL TRIAL: NCT07166224
Title: The Effect of Regular Home Use of Dual-light Antibacterial Photodynamic Therapy (aPDT) or the Use of a Powered Toothbrush in Older Individuals With Periodontitis and Mild Cognitive Impairment: a Randomized Controlled Trial.
Brief Title: The Effect of Regular Home Use of Dual-light Antibacterial Photodynamic Therapy (aPDT) or the Use of a Powered Toothbrush in Older Individuals With Periodontitis and Mild Cognitive Impairment.
Acronym: e-DENT II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blekinge Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BTH-6.1.1-0172-2025
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Diseases; Oral Halitosis
Keywords: Mild Cognitive Impairment; Oral health; Quality of life; Powered toothbrush
MeSH Terms: conditions — Periodontal Diseases; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: RCT-study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Partisipants with Lumoral Dual-Light aPDT + Manual Toothbrush (Experimental)
  Interventions: Device: Dual-Light aPDT Treatment - Lumoral
- Partisipants with Oral-B iO Powered Toothbrush (Experimental)
  Interventions: Device: Oral-B Powered toothbrush
- Control Group (No Intervention)

INTERVENTIONS:
Device: Oral-B Powered toothbrush — Intervention Group B:
  Participants receive standardized oral hygiene instructions and use an Oral-B iO powered toothbrush during the test period.
  The Oral-B iO is an advanced powered toothbrush that combines oscillating-rotating and micro-vibrating bristle movements with real-time feedback technology. It is CE-marked for home use and designed to improve plaque removal and overall oral hygiene compared to manual toothbrushing. The device incorporates pressure sensors and guided brushing modes to support optimal brushing technique and patient adherence, which may contribute to improved periodontal outcomes.
  Arms: Partisipants with Oral-B iO Powered Toothbrush
Device: Dual-Light aPDT Treatment - Lumoral — Intervention Group A:
  Participants receive standardized oral hygiene instructions and use only a manual toothbrush during the test period, with the addition of an adjunctive antimicrobial photodynamic therapy (aPDT) device (Lumoral®).
  The Lumoral® treatment device is a CE-marked antibacterial device intended for home use. It is designed to support the treatment and prevention of oral diseases caused by bacterial biofilms. The device functions by emitting light at a specific wavelength, which activates a CE-marked photosensitizing mouthrinse, Lumorinse®. This light-activated process enhances antibacterial efficacy, targeting pathogenic microorganisms in the oral cavity and supporting improved oral hygiene outcomes.
  Arms: Partisipants with Lumoral Dual-Light aPDT + Manual Toothbrush

SUMMARY:
Objective:

To compare three different oral hygiene regimens regarding plaque index (PI), bleeding on probing (BOP), the number of deepened periodontal pockets ≥4 mm (PPD), oral halitosis, and changes in oral health-related quality of life (OHRQoL) in an older population with periodontitis stage I-III and mild cognitive impairment.

1. Are there improvements in plaque index (PI), number of bleeding on probing (BOP) sites, number of probing depths (PPD), and intraoral halitosis in the two test groups compared to the control group?
2. Do the study interventions affect oral health-related quality of life in older adults with periodontitis and mild cognitive impairment?

Study design:

Type: Randomized controlled trial Duration: 6 months per participant, 2 years in total for data collection Participants: 90 participants divided into Intervention and Control groups

Intervention Group A (Lumoral Dual-Light aPDT + Manual Toothbrush) Standardized oral hygiene instructions and the use of a manual toothbrush during the test period, with an adjunctive aPDT device (Lumoral®).

Intervention Group B (Oral-B iO Powered Toothbrush) Standardized oral hygiene instructions and the use of an Oral-B iO powered toothbrush during the test period.

Control Group Standardized oral hygiene instructions and the use of a manual TePe Select extra soft toothbrush during the test period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥60 years
* ≥15 teeth
* Diagnosed periodontitis stage I-III
* MMSE score between 22-28
* Able to provide informed consent

Exclusion Criteria:

* Antibiotic use (within 3 months)
* Lumoral use within 3 months
* Bisphosphonate medication
* Immunosuppressive drugs or radiation therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in the amount of dental plaque | Assessments will be conducted at baseline, at 3 months, and at 6 months.
  Assessment will be performed on all teeth at six sites per tooth. The plaque index (PI) will be reported as the percentage of sites with visible plaque, providing an estimate of the overall plaque accumulation on the teeth.
Change in the amount of gingival bleeding on probing | Assessments will be conducted at baseline, at 3 months, and at 6 months.
  A full-mouth assessment will be performed at six sites per tooth. Bleeding on probing (BOP) will be reported as the percentage of sites exhibiting bleeding.
Change in the number of periodontal pockets ≥4 mm in depth | Assessments will be conducted at baseline, at 3 months, and at 6 months.
  Pocket depth will be measured from the base of the pocket to the gingival margin at six sites per tooth. Probing pocket depths (PPD) of ≥4 mm will be recorded.
MMSE-test | Baseline
  An 11-item cognitive assessment covering five domains: orientation, registration, attention and calculation, recall, and language. The maximum possible score is 30, with a score of 23 or lower indicating cognitive impairment.
Change in the amount of VSCs in the exhaled air | Assessments will be conducted at baseline, at 3 months, and at 6 months.
  Volatile sulfur compounds (VSCs) in exhaled air will be measured using the OralChroma® device. The cutoff values are as follows: H₂S ≥112 ppb, CH₃SH ≥26 ppb, and (CH₃)₂S ≥8 ppb.
Change in values for the oral health related quality of life instrument OHIP-14 | Assessments will be conducted from baseline to 6 months.
  Oral health-related quality of life will be assessed using the OHIP-14 (Oral Health Impact Profile-14) instrument. Scores range from 0 to 56, with lower scores indicating better oral health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Blekinge Tekniska Högskola, Karlskrona, Blekinge County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The trial protocol and the datasets used and analyzed during the current study are available upon reasonable request.
Supporting Information: Study Protocol
Access Criteria: The trial protocol and the datasets used and analyzed during the current study are available upon reasonable request.